CLINICAL TRIAL: NCT00142194
Title: Markers of Oxidative Stress Present in Blood in Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Samuel C. Dudley, Jr., Principal Investigator, Emory University
Other Study IDs: 476-2005
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation; Inflammation; Atrial Flutter
Keywords: Atrial Fibrillation; Oxidative stress; Cardiology
MeSH Terms: conditions — Atrial Fibrillation; Inflammation; Atrial Flutter

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Atrial fibrillation is an abnormal heart beat that starts in the upper parts of the heart and can cause stroke or death, if untreated. In general, treatments are not very effective, with frequent relapses of the abnormal heart beats. One explanation for the high relapse rate is that the treatments might not address the underlying cause of atrial fibrillation. Recently, the investigators have found that atrial fibrillation is associated with increased oxidative stress. This is a condition where abnormal oxygen forms are produced. These forms harm the cells of the heart, causing them to beat abnormally. The investigators have found increased oxidative stress in pig and mouse models of atrial fibrillation. They would like to see if oxidative stress is present in humans with atrial fibrillation. In this study, they will compare blood markers of oxidative stress between patients with and without atrial fibrillation. It is the expectation that participants with atrial fibrillation will have more abnormal blood markers of atrial fibrillation. This study requires participants to visit their doctors, undergo a history and physical examination, and give blood only once.

DETAILED DESCRIPTION:
Atrial fibrillation is an abnormal heart beat that starts in the upper parts of the heart and can cause stroke or death, if untreated. In general, treatments are not very effective with frequent relapses of the abnormal heart beats. One explanation for the high relapse rate is that the treatments might not address the underlying cause of atrial fibrillation.

Recently, we have found that atrial fibrillation is associated with increased oxidative stress in a particular part of the top parts of the heart, the left atrial appendage (LAA). Oxidative stress is a condition where abnormal oxygen forms are produced. These forms harm the cells of the heart, causing them to beat abnormally. Also, the inside of the heart becomes sticky and more likely to form blood clots. These clots, when they travel to the head, are thought to be the main cause of stroke in this condition. We have found increased oxidative stress and increased evidence of blood clotting in pig and mouse models of atrial fibrillation. We would like to see if these same findings are present in the human LAA.

In this study, we will compare blood and tissue markers of oxidative stress between patients with and without atrial fibrillation who are scheduled to undergo cardiac surgery. It is the expectation that participants with atrial fibrillation will have more abnormal markers of atrial fibrillation. This study requires participants to be seen during their routine preoperative visit, undergo a history and physical examination, give blood only once, and allow use of their discarded LAA. This tissue is routinely removed at surgery because its removal is thought to reduce the risk of stroke in patients who develop atrial fibrillation after the surgery. This happens in up to 50% of patients, thus providing the desire to remove the LAA.

ELIGIBILITY:
Inclusion Criteria:

* Cases must have atrial fibrillation documented on electrocardiographic recordings at the time of enrollment.

Exclusion Criteria:

* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years with or without permanent or persistent atrial fibrillation.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation (irregular heart beat coming from the upper chamber of the heart). To look at the differences between people who have irregular heart beats compared to those who do not have irregular beats. Study may last up until one year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Samuel C Dudley, M.D., Ph.D., Principal Investigator — Veterans Administration/Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Crawford Long Hospital, Atlanta, Georgia

REFERENCES:
- [Result] Neuman RB, Bloom HL, Shukrullah I, Darrow LA, Kleinbaum D, Jones DP, Dudley SC Jr. Oxidative stress markers are associated with persistent atrial fibrillation. Clin Chem. 2007 Sep;53(9):1652-7. doi: 10.1373/clinchem.2006.083923. Epub 2007 Jun 28. PMID 17599958